CLINICAL TRIAL: NCT05302674
Title: Short- and Long-term Health Consequences of Workers During Consecutive Days of Heat Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005847
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Heat Stress; Fatigue
MeSH Terms: conditions — Heat Stress Disorders; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hot Dry (Experimental): The participant will complete four hours of work at a 45:15 work rest cycle in a 98°F (36.7°C) and 20% relative humidity environment.
  Interventions: Other: Hot Dry

INTERVENTIONS:
Other: Hot Dry — 98°F (36.7°C) and 20% relative humidity environment

SUMMARY:
The purpose of this study is to measure fatigue and indicators of acute kidney injury during consecutive days of work in a hot environment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Regularly completes aerobic exercise at least 60 min per week

Exclusion Criteria:

* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* Hypertensive or tachycardic during the screening visit (Systolic Blood Pressure > 139 mmHg, Diastolic Blood Pressure > 89 mmHg, heart rate > 100 bpm)
* Current tobacco or nicotine use or previous regular use within the past 2 years
* Current or previous musculoskeletal injury limiting physical activity
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, beta blockers, diuretics, psychotropics, etc.)
* A positive pregnancy test at any point during the study or currently breastfeeding
* Study physician discretion based on any other medical condition or medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in fatigue | Hour 4
  Fatigue will be measured using accelerometry, with the primary variable being jerk, the smoothness or unevenness of movement.
Biomarkers of acute kidney injury | Hour 4
  Tissue inhibitor of metalloproteinase 2 (TIMP-2) and insulin-like growth factor binding protein 7 (IGFBP7) are biomarkers that have the potential for early prediction of acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Riana R Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Center for Research and Education in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to share individual participant data with other researchers. Aggregate results will be shared via publications and/or presentations.